CLINICAL TRIAL: NCT02283008
Title: Evaluating the Efficacy of 2 Different Educational Strategies for Improving and Maintaining Inhaler Technique
Brief Title: Inhaler Technique Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northampton General Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Steven Hickey, Respiratory Nurse Specialist, Northampton General Hospital NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRAS Project ID: 153018
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Asthma Chronic; Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): This arm will receive standard care which involves informal education on how to use metered dose inhalers
- Structured education (Active Comparator): This arm will receive structured education on the use of inhalers. At 6 weeks post education inhaler technique will be re-assessed. Participants who fail to achieve a set level of competence may be chosen for semi structured interview.
  Interventions: Behavioral: Assessment of inhaler technique pre and 6 weeks post training

INTERVENTIONS:
Behavioral: Assessment of inhaler technique pre and 6 weeks post training — Assessment of inhaler technique on day one. Education package and training on inhaler use at week 2. Final assessment to establish maintenance of inhaler competence at week 8
  Arms: Structured education

SUMMARY:
The evidence for poor inhaler technique is both well established and observed worldwide. What is unclear from the evidence is why individuals demonstrate poor technique, despite the majority admitting to having previously had instruction on inhaler technique. The primary research question is 'Will there be a difference between post education inhaler technique scores when comparing structured education against informal education?'

To try and establish why individuals use inhalers incorrectly a semi structured interview is proposed

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be anybody whose regular treatment requires inhaled medication. They will be included regardless of age, disease, inhaler device used or cognition.

Exclusion Criteria:

* The only exclusion criteria will be if a willing participant is not on an inhaler of any type.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Inhaler technique scores will be compared at 6 weeks post inhaler technique education. The proportion achieving proficiency will be compared between those recieving usual care and those recieving structured care. | 6 weeks per cohort